CLINICAL TRIAL: NCT00790855
Title: Phase I-II Study of Bendamustine in Patients With Acute Leukemia and High-Risk Myelodysplastic Syndrome (MDS)
Brief Title: Bendamustine in Acute Leukemia and MDS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Response
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0634
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Acute Lymphoblastic Leukemia; Chronic Myeloid Leukemia
Keywords: Bendamustine; Acute Leukemia; Leukemia; Acute myeloid leukemia; Myelodysplastic Syndrome; Acute lymphoblastic leukemia; Chronic myeloid leukemia; MDS; ALL; AML; CML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bendamustine (Experimental): Starting dose 50 mg/m^2 intravenously over 2 hours twice on Days 1-4 of every 4 week study cycle.
  Interventions: Drug: Bendamustine

INTERVENTIONS:
Drug: Bendamustine — Starting dose of 50 mg/m^2 through a needle or catheter in vein over 2 hours twice on Days 1-4 of every 4 week study cycle. A new study cycle may begin when blood cell counts have returned to an appropriate level or a new study cycle may begun earlier if disease gets worse or does not improve.
  Other Names: Treanda®; Bendamustine Hydrochloride; Bendamustine HCI; CEP-18083; SDX-105

SUMMARY:
The goal of the Phase I part of this clinical research study is to find the highest safe dose of bendamustine that can be given to patients with acute myelogenous leukemia (AML), Acute lymphoblastic leukemia (ALL), Chronic myelogenous (or myeloid) leukemia (CML) in blastic phase, Chronic Myelomonocytic Leukemia (CMML), and myelodysplastic syndromes (MDS).

The goal of the Phase II part of this clinical research study is to learn if bendamustine can help to control AML, ALL and MDS. The safety of this drug will continue to be studied.

DETAILED DESCRIPTION:
The Study Drug:

Bendamustine is designed to damage and destroy the DNA of cancer cells.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you joined this study. Up to 60 participants will be enrolled in the Phase I portion of the study, and up to 3 groups of 31 participants will be enrolled in Phase II.

If you are enrolled in the Phase I portion, the dose of bendamustine you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of bendamustine. Each new group will receive a higher dose of bendamustine than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of bendamustine is found.

If you are enrolled in the Phase II portion, you will receive bendamustine at the highest dose that was tolerated in the Phase I portion.

Study Drug Administration:

You will receive bendamustine through a needle or catheter in your vein over 2 hours twice on Days 1-4 of every 4 week study cycle. You will begin a new study cycle when your blood cell counts have returned to an appropriate level. You may begin a new study cycle earlier if your disease gets worse or does not improve.

Study Visits:

Blood (about 2 tablespoons) will be drawn for routine tests every 3-7 days during Cycle 1, and then every 1-2 weeks during all other cycles.

A bone marrow aspirate will be performed to check the status of the disease after Cycle 1 and every 3-4 Cycles thereafter, or as needed to document response.

Length of Study:

You may remain on study for as long as you are benefitting. You will be taken off study early if the disease gets worse or intolerable side effects occur.

This is an investigational study. Bendamustine is not FDA approved or commercially available in the United States. At this time, bendamustine is only being used in research.

Up to 153 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be 16 years of age or older.
2. Patients must have relapsed/refractory leukemias for which no standard therapies are anticipated to result in a durable remission (longer than 3 months). Patients with poor-risk myelodysplasia (MDS) [i.e. refractory anemia with excess blasts (RAEB-1 or RAEB-2) by World Health Organization (WHO) classification] and chronic myelomonocytic leukemia (CMML) are also candidates for this protocol. Relapsed/refractory leukemias include acute myeloid leukemia (AML), acute lymphocytic leukemia (ALL), or chronic myelogenous leukemia (CML) in blastic phase.
3. Continued from #2: Elderly patients with AML who are not eligible for frontline standard therapy, or who refuse to be treated with intensive chemotherapy, may be eligible. The phase II portion of the study will enroll patients with AML, MDS, and ALL. Patients with CML and CMML will not participate in the phase II portion of the study. Patients who are being considered for stem cell transplant are also eligible for this protocol.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-3.
5. Women of child-bearing potential (i.e., woman has not been naturally postmenopausal for at least 24 consecutive months or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative serum or urine pregnancy test within 2 weeks prior to beginning treatment on this trial. Sexually active men must also use acceptable contraceptive methods for the duration of time on study. Men and women must maintain effective contraception until 4 weeks after the last dose of drug is administered.
6. Must be able and willing to give written informed consent.
7. In the absence of rapidly progressing disease, the interval from prior treatment to time of study drug administration should be at least 2 weeks for cytotoxic agents, or at least 5 half-lives for noncytotoxic agents. If the patient is on hydroxyurea to control peripheral blood leukemic cell counts, the patient must be off hydroxyurea for at least 24 hours before initiation of treatment on this protocol. Persistent clinically significant toxicities (any grade 2 or worse toxicities, non-hematologic or hematologic) from prior chemotherapy must not be greater than Grade 1.
8. Patients must have the following clinical laboratory values unless considered due to leukemic organ involvement: 1) Serum creatinine </= 2.0 mg/dl; 2) Total bilirubin </= 1.5 times the upper limit of normal unless considered due to Gilbert's syndrome; 3) Alanine aminotransferase (ALT), or aspartate aminotransferase (AST) </= 3 times the upper limit of normal unless considered due to organ leukemic involvement.
9. Patients with active Central Nervous System (CNS) disease are included and will be treated concurrently with intrathecal therapy.
10. Phase II Portion: All above criteria apply. After the phase I portion, patients eligibility will be for only 3 disease categories which will accrue in parallel: 1) AML, 2) MDS, and 3) ALL.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to uncontrolled infection (i.e. persistent fever, clinical deterioration), acute congestive heart failure and exacerbation, cardiac arrhythmia, chronic liver disease, or psychiatric illness/social situations that would limit compliance with study requirements.
2. Active heart disease including myocardial infarction within previous 3 months, unstable angina, arrhythmias not controlled by medication, or uncontrolled congestive heart failure. Patients with New York Heart Association (NYHA) class 3 or 4 are excluded.
3. Patients receiving any other standard or investigational treatment for their hematologic malignancy, except as permitted under Inclusion #9 above.
4. Pregnant or breast feeding females are excluded because the effects of bendamustine on a fetus or nursing child are unknown.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop M. Kantarjian, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Details: 11/6/2008 to 9/1/2010. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: Out of 27 participants registered, two were found ineligible and did not participate in the study.
Period: Overall Study
Arm/Group | Bendamustine
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bendamustine
Number analyzed (Participants) | 25
Age Continuous [Median (Full Range); unit: years] | 57 [22 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD is the highest dose level in which <2 patients of 6 develop first cycle dose limiting toxicity (DLT). MTD assessed during course 1 (4 week cycle), every 3-7 days.
Time Frame: During course 1 (4 week cycle)
Measure: Number; unit: mg/m^2
Groups:
- Bendamustine: Starting dose 50 mg/m^2 intravenously, over 2 hours twice on Days 1-4 of every 4 week study cycle, with dose escalation of 25 mg/m^2 for 3 levels.
Arm/Group | Bendamustine
Number analyzed (Participants) | 25
mg/m^2 | 75

2. Secondary Outcome: Number of Participants With a Response
Description: A complete response (CR) is defined as normalization of the bone marrow and peripheral blood counts with </= 5% marrow blasts in a normo-or hypercellular marrow, with a granulocyte count of >/= 10^9/L and a platelet count of >/=100 X 10^9/L. A partial response (PR) was defined as for CR, but with only >/=50% reduction of marrow blasts and to a range of 6%-25%. A marrow complete response was defined as a reduction of marrow blasts to </=5% but without recovery of peripheral counts.
Time Frame: 1 - 24 week cycles (up to 8 weeks)
Measure: Number; unit: participants
Groups:
- Bendamustine (75 mg/m^2): 75 mg/m^2 intravenously over 2 hours twice on Days 1-4 of every 4 week study cycle.
Arm/Group | Bendamustine (75 mg/m^2)
Number analyzed (Participants) | 25
participants
  Complete Response | 0
  Partial Response | 0
  Marrow Complete Response | 1

ADVERSE EVENTS:
Time Frame: 3 years 3 months
Arm/Group | Bendamustine
Serious Adverse Events (participants affected / at risk) | 3/25
Other Adverse Events (participants affected / at risk) | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine (N=25)
Death (General disorders) | 1 (1)
Seizures (Nervous system disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine (N=25)
Elevated Creatinine (Renal and urinary disorders) | 11 (11)
Nausea/Vomiting (Gastrointestinal disorders) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Liver function abnormality (Metabolism and nutrition disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No